CLINICAL TRIAL: NCT02326584
Title: A Phase 1b Dose-escalation Study of SGN-CD33A in Combination With Standard-of-care for Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Safety Study of SGN-CD33A in Combination With Standard-of-care in Patients With AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN33A-002
Record Dates: First submitted 2014-12-18; First posted 2014-12-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia; Acute Myelogenous Leukemia
Keywords: Acute Myeloid Leukemia; Antibody-Drug Conjugate; CD33 Antigen; Drug Therapy; Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Neoadjuvant Therapy; vadastuximab talirine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Induction with SGN-CD33A (Experimental): 7+3 (Standard dose cytarabine for induction and daunorubicin) + SGN-CD33A
  Interventions: Drug: Standard dose cytarabine for induction; Drug: SGN-CD33A; Drug: Daunorubicin
- Consolidation with SGN-CD33A (Experimental): High dose cytarabine for consolidation + SGN-CD33A (28-day cycles)
  Interventions: Drug: SGN-CD33A; Drug: High dose cytarabine for consolidation
- SGN-CD33A Maintenance (Experimental): SGN-CD33A Monotherapy (42-day cycles)
  Interventions: Drug: SGN-CD33A
- Induction and Consolidation with SGN-CD33A (Experimental): 7+3 (standard dose cytarabine for induction and daunorubicin) + SGN-CD33A and High dose cytarabine for consolidation + SGN-CD33A
  Interventions: Drug: Standard dose cytarabine for induction; Drug: SGN-CD33A; Drug: Daunorubicin; Drug: High dose cytarabine for consolidation

INTERVENTIONS:
Drug: Standard dose cytarabine for induction — 100 mg/m2/day Days 1-7
  Arms: Induction and Consolidation with SGN-CD33A; Induction with SGN-CD33A
Drug: SGN-CD33A — Given intravenously Day 1 or Days 1 and 4 of each cycle
  Other Names: vadastuximab talirine
Drug: Daunorubicin — 60 mg/m2/day Days 1-3
  Arms: Induction and Consolidation with SGN-CD33A; Induction with SGN-CD33A
Drug: High dose cytarabine for consolidation — 3g/m2 on Days 1, 3, and 5 of each cycle
  Arms: Consolidation with SGN-CD33A; Induction and Consolidation with SGN-CD33A

SUMMARY:
This study will examine the safety profile of vadastuximab talirine (SGN-CD33A) by itself (monotherapy) or in combination with other standard treatments. The main purpose of this study is to find the best dose and schedule for SGN-CD33A when given in combination with standard induction treatment, in combination with standard consolidation treatment, or by itself for maintenance treatment. This will be determined by observing the dose-limiting toxicities (the side effects that prevent further increases in dose) of SGN-CD33A. In addition, the pharmacokinetic profile and anti-leukemic activity of the study treatment will be assessed.

DETAILED DESCRIPTION:
The study will be conducted in the following distinct parts:

Part A: Induction dose escalation - 7+3 combined with SGN-CD33A (Day 1 and Day 4 dosing)

Part B: Consolidation dose escalation - consolidation combined with SGN-CD33A; up to 4 cycles of consolidation therapy will be administered after SGN-CD33A (Day 1 of each cycle).

Part C: Maintenance - SGN-CD33A Monotherapy; Up to 24 patients with and up to 24 patient without prior allogeneic stem cell transplant will be treated with SGN-CD33A. Both arms will enroll simultaneously. SGN-CD33A will be administered on Day 1 of each 6-week cycle for up to 8 cycles.

Part D: Induction plus consolidation - induction/consolidation combined with SGN-CD33A; patients who achieve a CR/CRi (with or without a second induction) will receive up to 4 cycles of consolidation therapy administered after SGN-CD33A (Day 1 of each cycle).

Part E: Induction dose escalation - 7+3 combined with SGN-CD33A (Day 1 dosing)

ELIGIBILITY:
Inclusion Criteria:

* All subtypes of Acute Myeloid leukemia (except for acute promyelocytic leukemia)
* Eastern Cooperative Oncology Group status of 0 or 1
* Adequate baseline renal and hepatic function
* Central venous access
* Part specific requirements: eligible to receive induction; achieved CR/CRi with standard induction and eligible to receive consolidation; in CR with documented blood count recovery for maintenance

Exclusion Criteria:

* Previous treatment for MDS or MPN for dose escalation cohorts
* Inadequate lung function
* Inadequate heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-30 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose
Incidence of laboratory abnormalities | Through 1 month following last dose
Incidence of dose-limiting toxicity (DLT) | Through 1 month following last dose

SECONDARY OUTCOMES:
Complete remission (CR) rate at the end of induction | Through 1 month following last dose
Leukemia-free survival | Up to approximately 3 years
Overall survival | Up to approximately 3 years
Blood concentrations of SGN-CD33A and metabolites | Up to approximately 3 years
Incidence of antitherapeutic antibodies (ATA) | Up to approximately 3 years
Rate of minimal residual disease (MRD) clearance | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Feldman, MD, Study Director — Seagen Inc.
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, The, Cleveland, Ohio
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington